CLINICAL TRIAL: NCT01724333
Title: International Validation and Testing of a Supplementary Questionnaire Module for Assessment of Oral and Dental Health in Cancer; the QLQ-OH17
Brief Title: International Validation of the QLQ-OH17 for Oral Health
Acronym: QLQ-OH17
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Principal Investigator, Marianne Jensen Hjermstad, Senior researcher, Oslo University Hospital
Other Study IDs: 2012/1390REK; EORTC-SG2012 (Other Grant/Funding Number: EORTC)
Record Dates: First submitted 2012-11-02; First posted 2012-11-09 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Quality of Life; Adverse Effects; Late Effects; Cancer; Xerostomia
Keywords: EORTC QLQ-C30; Oral health; Quality of life; Questionnaires; Patient reported; outcomes
MeSH Terms: conditions — Neoplasms; Xerostomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Group 1- in active treatment: Questionnaires only
- Group 2 - 2-6 months post-treatment: Questionnaires only
- Group 3 - 6 mos-3yrs post-treatment: Questionnaires only
- Group 4 - Palliative treatment: Questionnaires only
- Group 5 - Referred to dentist/oral team: Questionnaires only

SUMMARY:
Assessment of oral and dental problems is seldom routine in clinical oncology, despite the potential negative impact of these problems on nutritional status, social function and quality of life (QoL). A brief, assessment tool for oral/dental health and related QoL-issues to improve symptom management has been requested. The present study will be conducted on behalf of and with support from the European Organisation for Research and Treatment of Cancer - (EORTC) Quality of Life Group (QLG). The study represents phase IV, the final step, in the development of an international, symptom specific questionnaire module, focusing on oral and dental problems in relation to cancer and its treatment. Phase I-III of this stepwise development process was conducted from 2008 to 2011, as an international collaboration and conducted according to the guidelines for module development set forth by the EORTC QLG. The resulting module, the QLQ-OH17, is now subject to an international field testing and validation study as described in this project description.

The present version of the QLQ-OH17 consists of 17 items conceptualized into four multi-item scales (pain/discomfort, xerostomia, eating and information) and three single items related to use of dentures and future worries. The aim of the present study is to conduct phase IV; an international field study to confirm the psychometric properties of the QLQ-OH17

DETAILED DESCRIPTION:
The EORTC guidelines will be strictly followed also in phase IV of the module development. Eligible patients will be contacted by the local study coordinator or a study nurse and informed about the study. After having provided written informed consent, they will be presented with the following two questionnaires for self-report of general symptoms, specific dental and oral symptoms, and quality of life issues; the EORTC QLQ-C30 and the QLQ-OH17. In addition to these two, a short debriefing interview will be conducted by study coordinator / study nurse for assessment of feasibility and patients' opinion about the questionnaires.

The case report form (CRF) on medical and demographic data will be completed by the study coordinator / study nurse before or after the patients have completed their part.

A subset of the patients will be assessed twice, as examination of test - retest reliability is important in phase IV of the development process.

ELIGIBILITY:
Inclusion Criteria

* Patients with a verified cancer diagnosis other than basal cell carcinoma, incl. H&N cancer
* Sufficient language ability to understand and complete the questionnaires without assistance
* No obvious cognitive impairments, as judged by the study coordinator upon inclusion
* Age 18 years or above
* Provision of written informed consent
* No participation in another trial or study possibly interfering with the present study

Exclusion Criteria:

* Patients being diagnosed with basal cell carcinoma
* Patients who have been included in Phase I-III of the module development
* Patients who are in the terminal phase of cancer
* Patients who are unable to participate in the interviews do to obvious cognitive impairment, psychological disturbance or language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An international, cross-cultural sample of cancer patients with different diagnoses in different phases of treatment
Sampling Method: Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Oral morbidity | Up to two years
  The study aims to validate a questionnaire for assessment of oral morbidity, oral health , and quality of life in relation to cancer treatment. Specific outcomes are prevalence of patients with moderate to severe oral morbidity due to cancer treatment (mucositis,stomatitis, taste change, decayed /loose teeth, osteoradionecrosis, ulcers), to investigate if the severity varies with certain background variables , for example, diagnostic group, age, sex, stage of disease, type of treatment, and to investigate the discriminant validity, reliability and responsiveness of the specific items in patient subgroups

SECONDARY OUTCOMES:
Quality of life | Up to two years
  The questionnaire module that is subject to testing of psychometric properties, will be used together with a well-validated quality of life questionnaire, to investigate if oral morbidity affects overall quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Marianne J Hjermstad, PhD, Principal Investigator — Oslo University Hospital
Locations (14):
- University of Metz, Metz, France
- Germany (2):
  - University of Leipzig, Leipzig
  - Johannes Gutenberg University Mainz, Mainz
- University of Athens, Athens, Greece
- Tel-Aviv University, Tel Aviv, Israel
- Istituto Nazionale Tumori "Fondazione G. Pascale"- IRCCS,, Naples, Italy
- Netherlands (2):
  - Academic Centre for Dentistry Amsterdam, Amsterdam
  - VU University Medical Center, Amsterdam
- Norway (2):
  - Oslo University Hospital, Oslo
  - University of Oslo, Oslo
- Poland (2):
  - J. Dietl Specialistic Hospital,, Krakow
  - Jagiellonian University Medical College, Krakow
- Karolinska University Hospital, Stockholm, Sweden
- University of Leeds, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Phase III and Phase IV reports approved by the EORTC Quality of Life Group Executive Committee. First publication in Eur J Cancer. 2012 Sep;48(14):2203-11. doi: 10.1016/j.ejca.2012.04.003. Second publication accepted for publication in Supp Care Cancer, April 2016

REFERENCES:
- [Background] Hjermstad MJ, Bergenmar M, Bjordal K, Fisher SE, Hofmeister D, Montel S, Nicolatou-Galitis O, Pinto M, Raber-Durlacher J, Singer S, Tomaszewska IM, Tomaszewski KA, Verdonck-de Leeuw I, Yarom N, Winstanley JB, Herlofson BB; EORTC QoL Group. International field testing of the psychometric properties of an EORTC quality of life module for oral health: the EORTC QLQ-OH15. Support Care Cancer. 2016 Sep;24(9):3915-24. doi: 10.1007/s00520-016-3216-0. Epub 2016 Apr 25. PMID 27113466
- [Result] Hjermstad MJ, Bergenmar M, Fisher SE, Montel S, Nicolatou-Galitis O, Raber-Durlacher J, Singer S, Verdonck-de Leeuw I, Weis J, Yarom N, Herlofson BB. The EORTC QLQ-OH17: a supplementary module to the EORTC QLQ-C30 for assessment of oral health and quality of life in cancer patients. Eur J Cancer. 2012 Sep;48(14):2203-11. doi: 10.1016/j.ejca.2012.04.003. Epub 2012 May 8. PMID 22572480
- [Derived] Johns SA, Brown LF, Beck-Coon K, Talib TL, Monahan PO, Giesler RB, Tong Y, Wilhelm L, Carpenter JS, Von Ah D, Wagner CD, de Groot M, Schmidt K, Monceski D, Danh M, Alyea JM, Miller KD, Kroenke K. Randomized controlled pilot trial of mindfulness-based stress reduction compared to psychoeducational support for persistently fatigued breast and colorectal cancer survivors. Support Care Cancer. 2016 Oct;24(10):4085-96. doi: 10.1007/s00520-016-3220-4. Epub 2016 May 17. PMID 27189614